CLINICAL TRIAL: NCT02347228
Title: A Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Clinical Activity of OB318 in Patients With Advanced Solid Malignancies
Brief Title: Evaluate Safety, Tolerability, PK, Preliminary Clinical Activity of OB318 in Patients With Advanced Solid Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB318CLCT01
Record Dates: First submitted 2014-12-25; First posted 2015-01-27 (Estimated); Last update posted 2024-01-26 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Malignancies
Keywords: OB318; Advanced Solid Malignancies; Antrodia cinnamomea; Antrodia camphorata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OB318 capsule (Experimental)
  Interventions: Drug: OB318 capsule

INTERVENTIONS:
Drug: OB318 capsule — Oral qd, at least 30 minutes before breakfast

SUMMARY:
The objectives of this Phase I study are to determine the maximum tolerable dose (MTD) and to evaluate pharmacokinetics (PK), safety/ tolerability and preliminary efficacy of OB318 in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients of age ≥20 years
2. Pathologically or cytologically confirmed advanced solid tumors for which standard therapy proven to provide clinical benefit does not exist or is no longer effective; the diagnosis of hepatocellular carcinoma (HCC) made according to the imaging specified in the American Association for the Study of Liver Diseases (AASLD) 2018 is acceptable.
3. Evaluable disease, either at least one measurable untreated target lesion on imaging by RECIST 1.1 (Response Evaluation Criteria in Solid Tumors) criteria or measurable by informative tumor marker(s).
4. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2.
5. Life expectancy ≥ 3 months.
6. If history of brain metastases treated with radiation therapy, radiation therapy is required to be completed at least 3 months prior to enrolment and metastasis achieve stable disease (SD) since radiation completion.
7. Must have recovered from toxicities of previous anti-cancer treatments to NCI-CTCAE grade 1 or lower, except for alopecia.
8. Laboratory values at screening of:

   * Absolute neutrophil count ≥ 1,500 /mm3;
   * Platelets ≥ 75,000 /mm3;
   * Hemoglobin (Hb) ≥ 8.5 g/dL;
   * Total bilirubin ≤2.0 mg/dL;
   * AST (SGOT) ≤ 3 × ULN (upper limit of normal);
   * ALT (SGPT) ≤ 3 × ULN;
   * Serum creatinine ≤1.5 mg/dL or a measured creatinine clearance ≥ 60 mL/min.
9. Patients with primary liver cancer or hepatic metastasis are eligible to enroll, provided that, at screening, the following criteria are met:

   * Total bilirubin ≤2.0 mg/dL;
   * AST and ALT ≤ 5 × ULN;
   * Child-Pugh Class A;
   * Patients with a history of esophageal bleeding have varices that have been sclerosed or banded and no bleeding episodes have occurred during the prior 6 months.
10. Female patients must be either of non-childbearing potential, i.e. surgically sterilized or one year post-menopausal; or, if of childbearing potential, confirmed not pregnant at screening and must use adequate contraceptive precautions (as per investigator) during the entire treatment period of this study and for 6 months after exiting from the study.
11. Male patients with female partners of childbearing potential must be willing to use a reliable form of contraception (as per investigator), from screening until 6 months after exiting from the study.
12. Given signed and dated written informed consent and willing/able to comply with all protocol required visits/procedures

Exclusion Criteria:

1. Primary major surgery < 4 weeks prior to the planned first study treatment day.
2. Lactating or pregnant women or plans to be become pregnant.
3. Except for alopecia, any drug-related AE from any previous treatments not recovered to grade 1 or less prior to the planned first study treatment day.
4. With active systemic infections, active and clinically significant cardiac diseases, active gastrointestinal diseases, active pulmonary diseases, or medical conditions that may significantly affect adequate absorption of investigational product, eg., bad nutrition, proteinuria, etc..
5. Previous malignancy, except for basal-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was treated with curative intent more than 2 years prior to study entry.
6. Known allergic to OB318 or its formulation excipients.
7. History of autoimmune disease.
8. Taking anti-coagulant or anti-platelet drugs (eg aspirin, Coumadin, ginko, clopidogrel).
9. Use of any investigational agents or non-registered product within 4 weeks of baseline.
10. Known human immunodeficiency virus (HIV) positivity.
11. With conditions, judged by the investigator, as unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) of OB318 | 28 days
  NOTE: DLT is defined as any grade 3 or above toxicity by NCI-CTCAE version 4.03, as determined by the investigator and sponsor, to be at least possibly related in causality to the administered investigational product OB318 and will be observed during the 4 weeks of treatment for patients in the dose escalation phase.
Maximum tolerated dose (MTD) of OB318 | 28 days
  NOTE:- MTD is defined as the prior dose level below the dose level at which 2/3 or 2/6 subjects suffer dose limiting toxicity (DLT) in the dose escalation phase

SECONDARY OUTCOMES:
Changes in laboratory safety tests (hematology, biochemistry, urinalysis) from baseline | up to 84 days
  Laboratory safety tests will be performed at screening, baseline, Day 14 and Day 28 for the dose escalation, and at the last follow-up visit. For the extension phase, lab tests will be done before each 28 days cycle.
Incidence of Adverse Events (AEs) | up to 84 days
Incidence of Serious Adverse events (SAEs) | up to 84 days
Incidence of toxicities ≥ grade 3, according to NCI-CTCAE version 4.03, related to OB318, during extension phase | up to 84 days
Characterization of toxicities ≥ grade 3, according to NCI-CTCAE version 4.03, related to OB318, during extension phase | up to 84 days
Changes in physical examination from baseline | up to 84 days
  Physical examination will be performed at screening, baseline, and Day 28 for the dose escalation, and at the last follow-up visit. For the extension phase, physical examination will be done at last day of each cycle.
Changes in vital signs from baseline | up to 84 days
  Vital signs will be performed at each study visit.
Changes from baseline in Electrocardiogram (ECG) results (QRS, QT, QTc, RR intervals) | up to 84 days
  Electrocardiogram (ECG) is conducted at screening, baseline, Day 14 and Day 28 for the dose escalation, and at the last follow-up visit. For the extension phase, ECG will be conducted at the same time.
Tumor response per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 at the end of the | up to 84 days
  Imaging for tumor assessment will be made at screening, at the end of the treatment for the dose escalation and at the end of Cycle 2 for the extension phase.
Pharmacokinetic parameters- Cmax | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- AUC from time zero to the last quantifiable concentration | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- AUC from time zero extrapolated to infinity | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters-CL/F | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters-Vz/F | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters-Tmax | Day 1 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Terminal elimination half-life | Day 1 and Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Terminal elimination rate constant | Day 1 and Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters-Ctrough | Day 27 and Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318 ; Day 7 and Day 14 of Cycle additionally for dose level 1 only
Pharmacokinetic parameters- Cmin,ss | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Cmax,ss | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Cavg,ss | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- AUC(0-24h) | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- CLss/F | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Vz,ss/F | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Tmax,ss | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- FI | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318
Pharmacokinetic parameters- Rac | Day 28 of Cycle 1 from the subjects with dose level 1, 2, 4, 6, 8, and 10 of OB318

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Ho, Principal Investigator — Tri-Service General Hospital
Locations (2):
- Taiwan (2):
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei